CLINICAL TRIAL: NCT05559333
Title: CLINICAL COMPARISON OF DIFFERENT GLASS IONOMER-BASED RESTORATIVES AND A BULK-FILL RESIN COMPOSITE IN CLASS I CAVITIES: A 48-MONTH RANDOMIZED SPLIT-MOUTH CONTROLLED TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ece Meral, assistant professor, Hacettepe University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KA-17057
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Class I Dental Caries
Keywords: glass ionomer cements; bioactive materials

STUDY DESIGN:
Intervention Model Description: randomized-split mouth clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- zirconomer (Active Comparator): zirconia reinforced glass ionomer cement
  Interventions: Procedure: class I restoration placement
- Equia Fil (Active Comparator): High viscosity glass ionomer cement
  Interventions: Procedure: class I restoration placement
- glass carbomer (Active Comparator): glass ionomer cement containing nano sized- carbonized particles.
  Interventions: Procedure: class I restoration placement
- Tetric-evo ceram bulk fill (Active Comparator): Bulk fill composite resin
  Interventions: Procedure: class I restoration placement

INTERVENTIONS:
Procedure: class I restoration placement — zirconomer, glass carbomer, glass ionomer and composite resin class I restorations were placed.

SUMMARY:
The aim of this study is to compare the clinical performances of high-viscosity glass ionomer (GI), glass carbomer (GC), zirconia-reinforced GI (ZIR), and bulk-fill (BF) composite resin restorations.For this purpose, two calibrated operators placed 128 restorations in 30 patients with a mean age of 21 years. The restorations will be evaluated by one examiner at baseline and at 6, 12, 18,24, and 48 months using the modified US Public Health Service criteria. The data will statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting 1) at least four single-surface occlusal caries on their posterior molar teeth (first and/or second molars); 2) teeth to be restored had to be vital and without pulpal or periodontal disease, pain, and preoperative sensitivity; 3) teeth should be in occlusion; and 4) must agree to come to follow-up appointments.

Exclusion Criteria:

* patients with 1) poor oral hygiene, serious health problems, and/or heavy bruxism; 2) partly erupted teeth; 3) absence of adjacent and antagonist teeth; 4) teeth with interproximal caries; and 5) inability to attend recalls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Retention Alpha for at least 90% of the restorations | 24 months
  The primary factor for determining the clinical performance of a restorative material is the retention rate. It represents the survival rates of the restorations after a period of time. According to ADA guidelines, a restorative material should show at leat 90% alpha retention rate after 18 months to be considered as clinically acceptable. The retention is assesed as alpha (retentive restoratation) or charlie (failed restoration). Clinical evaluation is performed to examine if the restoration is in place or has fallen.

SECONDARY OUTCOMES:
marginal adaptation score alpha | 24 months
  It represents the marginal integrity of the restorations. It is scored as alpha (perfect marginal adaptation), bravo (detectable marginal discrepency, clinically acceptable) or charlie (marginal crevice, clinically unacceptable). The examination of marginal adaptation is performed by clinical examination of the restoration with probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided